CLINICAL TRIAL: NCT02692729
Title: Transverse Supraumbilical Versus Pfannenstiel Incision For Cesarean Section in Morbid Obese Patients" A Single Blinded Randomized Controlled Trial"
Brief Title: Transverse Supraumbilical Versus Pfannenstiel Incision for Cesarean Section in Morbidly Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed El Kotb Abdel Fattah, dr. Ahmed Kotb, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STIP
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2016-07

CONDITIONS: Cesarean Section

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- supraumbilical transverse (Experimental): transverse Supraumbilical Incision, in which the skin incision is a straight transverse skin incision slightly higher than the Pfannenstiel (5- 6) cm. from the upper border of the symphysis pubis The high transverse incision facilitated access to the fascia of the rectus abdominalis. Above the panniculus, the fatty tissues are not particularly thick. A transverse opening of the aponeurosis and of the parietal peritoneum was done. Then the approach to the lower uterine segment was easy. A Ricard retractor was put in place.
  Interventions: Procedure: transverse supraumbilical
- pfannenstiel (Active Comparator): Pfannenstiel Incision, in which the skin incision is a transverse upward concavity, typically initiated two finger-breadths above the symphysis pubis and extended in the direction of the anterior superior iliac spine below and medial to it about (2 - 3 ) cm.
  Interventions: Procedure: pfannenstiel incision

INTERVENTIONS:
Procedure: transverse supraumbilical — transverse Supraumbilical Incision, in which the skin incision is a straight transverse skin incision slightly higher than the Pfannenstiel (5- 6) cm. from the upper border of the symphysis pubis The high transverse incision facilitated access to the fascia of the rectus abdominalis
  Arms: supraumbilical transverse
Procedure: pfannenstiel incision — Pfannenstiel Incision, in which the skin incision is a transverse upward concavity, typically initiated two finger-breadths above the symphysis pubis and extended in the direction of the anterior superior iliac spine below and medial to it about (2 - 3 ) cm.
  Arms: pfannenstiel

SUMMARY:
This study aims to evaluate the efficacy and safety of transverse supraumbilical incision over Pfannenstiel incision in performing cesarean section for morbid obese pregnant women.

DETAILED DESCRIPTION:
Research Question In Morbidly obese women undergoing cesarean section, is transverse supraumbilical incision superior to Pfannenstiel incision? Research Hypothesis Transverse supraumbilical incision is superior to Pfannenstiel incision in morbidly obese women undergoing cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* BMI more than 40 kg/m2
* women scheduled for CS

Exclusion Criteria:

* patients receiving steroids or anticoagulation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
occurence of surgical site infection | one week
  occurance of redness, hotness, pus discharge and exudation

SECONDARY OUTCOMES:
operative time in minutes | 2 hours
  from skin incision to closure of the skin
blood loss in milliliter | 2 hours
  volume of blood during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M kotb, MD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] AbdElhady RM, Hamid ASA, El Sayed HM, El Mekkawi SF, Elhossary HMAF, El Kotb AM. Randomized trial assessing transverse supraumbilical incisions for cesarean sections in morbid obese women with pannus. BMC Pregnancy Childbirth. 2025 Dec 18. doi: 10.1186/s12884-025-08530-y. Online ahead of print. PMID 41413498